CLINICAL TRIAL: NCT01407393
Title: Double-blind, Randomized, Placebo-controlled, Bicentric Clinical Investigation to Evaluate Safety and Efficacy of Glucosanol in Reducing Body Weight in Overweight and Obese Subjects
Brief Title: Safety and Efficacy of Glucosanol in Reducing Body Weight in Overweight and Obese Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INQ/K/003411
Record Dates: First submitted 2011-06-30; First posted 2011-08-02 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Overweight and Obesity
Keywords: overweight; obesity; weight loss; body fat; waste cirumference; satiety; appetite
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucosanol (Experimental): Glucosanol
  Interventions: Device: Glucosanol
- Placebo (Placebo Comparator): Placebo
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Glucosanol — 2 tablets 3x daily for 12 weeks
  Arms: Glucosanol
Device: Placebo — 2 tablets 3x daily for 12 weeks
  Arms: Placebo

SUMMARY:
Glucosanol™, the medical device to be investigated contains a proprietary plant extract that is a natural inhibitor of alpha-amylase and can reduce starch digestion.

The rationale for this study is to confirm that Glucosanol™ ingestion will reduce body weight. A double-blind, randomized, placebo-controlled design has been chosen to assess the efficacy and safety of Glucosanol™ in subjects who are overweight and mildly obese.

DETAILED DESCRIPTION:
Preparations that reduce absorption of calories from dietary carbohydrates could be decisively meaningful for the regulation of bodyweight or obesity. Hence, Glucosanol™ may be used as a tool for the treatment of obesity and weight management through reduced carbohydrate absorption.

The rationale for this study is to confirm that Glucosanol™ ingestion will reduce body weight. A double-blind, randomized, placebo-controlled design has been chosen to assess the efficacy and safety of Glucosanol™ in subjects who are overweight and mildly obese.

The specific hypotheses to be accepted or rejected by statistical data from the clinical investigation are beneficial effects of the device on weight loss (kg) and body fat content.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* BMI between 25 and 35
* Expressed desire for weight loss
* Accustomed to 3 main meals/day
* Consistent and stable body weight 3 months prior to study enrolment
* Commitment to avoid the use of other weight loss products during study
* Commitment to adhere to diet recommendation
* Females' agreement to use appropriate birth control methods during the active study period
* Subject declares in writing his/her consent to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

* Known sensitivity to the ingredients of the device
* History of Diabetes mellitus
* Fasting blood glucose >7 mmol/L
* History or clinical signs of endocrine disorders which may influence body weight (e.g., Cushing's disease, thyroid gland disorders)
* Clinically relevant excursions of safety parameter
* Current use of anti-depressants
* Presence of acute or chronic gastrointestinal disease (e.g., IBD, coeliac disease. pancreatitis)
* Uncontrolled hypertension (>160/110 mm Hg)
* Stenosis in the GI tract
* Bariatric surgery
* Abdominal surgery within the last 6 months prior to enrollment
* History of eating disorders such as bulimia, anorexia nervosa within the past 12 months
* Other serious organ or systemic diseases such as cancer
* Any medication that could influence GI functions such as antibiotics, laxatives, opioids, glucocorticoids, anticholinergics, or antidiarrheals (e.g., loperamide; must have stopped 1 months before study start)
* Pregnancy or nursing
* Any medication or use of products for the treatment of obesity
* More than 3 hours strenuous sport activity per week
* History of abuse of drugs, alcohol or medication
* Smoking cessation within 6 months prior to enrolment
* Inability to comply due to language difficulties
* Participation in similar studies or weight loss programs within 3 months prior to enrolment
* Participation in other studies within 4 weeks prior to enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  The primary endpoint of this randomized, double-blind, placebo-controlled bicen-tric study is to assess the weight loss effect of Glucosanol™ (kg), in combination with a weight loss program in overweight and obese subjects.

SECONDARY OUTCOMES:
Proportion body weight | 12 weeks
  To assess the efficacy of Glucosanol™ to increase the proportions of subjects who lose at least 3% and 5% of baseline body weight
waist circumference | 12 weeks
  Changes in waist circumference
hip circumference | 12 weeks
  Changes in hip circumference
waist-hip-ratio | 12 weeks
  Changes in waist-hip-ratio
BMI | 12 weeks
  Changes in BMI
body fat | 12 weeks
  Changes in body fat (% and kg) and fat free mass (kg)
hunger | 12 weeks
  Changes in hunger, eating, and food craving-related items from a Control of Eating Questionnaire
Global evaluation of feeling of satiety | 12 weeks
  This parameter will be assessed by a 4 points categorical scale
Global evaluation of the efficacy | 12 weeks
  This parameter will be assessed by a 4 points categorical scale
Global evaluation of safety | 12 weeks
  This will be assessed by both investigators and subjects by a 4 points categorical scale.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grube, MD, Principal Investigator
Locations (1):
- Barbara Grube, Berlin, Germany